CLINICAL TRIAL: NCT01458028
Title: A Parallel Group, Double-Blind Study to Evaluate the Effects of Age and Gender on the Single-Dose Pharmacokinetics of BAY85-3934, Tablet Formulation
Brief Title: Age and Gender Effects on the Pharmacokinetics of BAY85-3934
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14631
Record Dates: First submitted 2011-09-20; First posted 2011-10-24 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Anemia
Keywords: BAY85-3934; pharmacokinetics; age; gender
MeSH Terms: conditions — Anemia; Coitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: BAY85-3934
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY85-3934 — Single doses of 20 mg BAY85-3934 as tablet
  Arms: Arm 1
Drug: Placebo — Single dose of placebo tablet matching the 20 mg BAY85-3934 tablet
  Arms: Arm 2

SUMMARY:
Single dose study of BAY85-3934 compared to placebo in young/elderly male and female healthy subjects. The main focus of the study is to determine if the pharmacokinetics (drug levels in blood) of BAY85-3934 is similar or not in the four subject groups. Qualifying subjects will be dosed with a single tablet of BAY85-3934 (or placebo) and blood will be drawn over 4 days. The safety and tolerability of BAY85-3934 compared to placebo will also be evaluated over the 5 days of the study.

ELIGIBILITY:
Inclusion Criteria:

* No diagnosis of any specific disease or condition
* Subjects are expected to be in good general health for their respective age range
* Male or female gender
* Age subgroups: 1) 18 to 45 years (inclusive) and 2) 65 to 85 years (inclusive)
* Racial group: Caucasian

Exclusion Criteria:

* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal. This includes moderate and severe renal impairment (on dialysis or not), and moderate or severe hepatic disease.
* Clinically relevant findings in the physical examination

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration vs time curve from zero to infinity after single (first) dose of BAY85-3934 | Measured over 72 hours after dosing
Maximum drug concentration in plasma after single dose administration of BAY85-3934 | Measured over 72 hours after dosing
Safety and tolerability of BAY 85-3934 after single dose administration as determined by physical examination (changes from baseline) | Measured over 96 hours after dosing
Safety and tolerability of BAY 85-3934 after single dose administration as determined by adverse events monitoring (number of subjects with a specific event) | Measured over 96 hours after dosing
Safety and tolerability of BAY 85-3934 after single dose administration as determined by electrocardigram and and vital sign measurememnt (changes from baseline) | Measured over 72 hours after dosing
Safety and tolerability of BAY 85-3934 after single dose administration as determined by laboratory testing (changes from baseline) | Measured over 48 hours after dosing

SECONDARY OUTCOMES:
Pharmacodynamic effects on erythropoietin as the change from baseline at 48 hours | 48 hours post dose
Pharmacodynamic effects on reticulocytes as the change from baseline at 96 hours | 96 hours post dose
Pharmacodynamic effects on hemoglobin as the change from baseline at 48 hours | 48 hours post dose
Pharmacodynamic effects on hematocrit as the change from baseline at 96 hours | 96 hours post dose
Pharmacodynamic effects on vascular endothelial growth factor (VEGF) as the change from baseline at 96 hours | 96 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Fargo, North Dakota, United States